CLINICAL TRIAL: NCT00835588
Title: A Relative Bioavailability Study of Pantoprazole Sodium 40 mg DR Tablets Under Fasting Conditions
Brief Title: Pantoprazole Sodium 40 mg DR Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B036581
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pantoprazole (Experimental): Pantoprazole Sodium 40 mg DR Tablet (test) dosed in first period followed by Protonix® 40 mg DR Tablet (reference) dosed in second period
  Interventions: Drug: Pantoprazole Sodium 40 mg delayed-release tablets
- Protonix® (Active Comparator): Protonix 40 mg DR Tablet (reference) dosed in first period followed by Pantoprazole Sodium 40 mg DR Tablet (test) dosed in second period
  Interventions: Drug: PROTONIX® 40 mg delayed-release tablets.

INTERVENTIONS:
Drug: Pantoprazole Sodium 40 mg delayed-release tablets — 1 x 40 mg
  Arms: Pantoprazole
Drug: PROTONIX® 40 mg delayed-release tablets. — 1 x 40 mg
  Arms: Protonix®

SUMMARY:
The objective of this study is to compare the relative bioavailability of pantoprazole sodium 40 mg delayed-release tablets ( manufactured by TEVA Pharmaceuticals Industries, Ltd. and distributed by TEVA Pharmaceuticals USA) with that of PROTONIX® 40 mg delayed-released tablets (Wyeth-Ayerst) in Healthy, adult, non-smoking subjects under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* All subjects selected for this study will be non-smokers at least 18 years of age. Subjects will have a BMI(Body Mass Index) of 30 or less.

Exclusion Criteria:

* Subjects with a significant recent history of chronic alcohol consumption (past 2 years), drug addiction, or serious gastrointestinal, renal, hepatic or cardiovascular, disease, tuberculosis, epilepsy, asthma (past 5 years), diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are greater than 20% outside the normal range may be retested. If the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result not to be significant.
* Subjects who have a history of allergic responses to the class of drug being tested will be excluded from the study.
* All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at each dosing period check-in. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least thirty (30) days prior to the first dosing of the study will not be allowed to participate.
* Female subjects who are pregnant, breast-feeding, or who are likely to become pregnant during the study will not be allowed to participate. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (e.g. condom, IUD) of contraception during the course of the study (first dosing until last blood collection) or they will not be allowed to participate. Subjects who have used implanted or injected hormonal contraceptives anytime during the 180 days prior to study dosing or oral hormonal contraceptives with in 14 days of dosing will not be allowed to participate.
* All female subjects will be screened for pregnancy at check-in each study period. Subjects with positive or inconclusive results will be withdrawn from the study.
* Subjects who do no tolerate venipuncture will not be allowed to participate.
* Subjects who use tobacco in any form will not be eligible to participate in the study. Three months abstinence is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-12; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Herrmann, M.D.; Ph.D, Principal Investigator — Cetero Research, San Antonio
Locations (2):
- United States (2):
  - Gateway Medical Research, Inc., Saint Charles, Missouri
  - Bioassay Laboratory, Inc., Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Pantoprazole (Test) First: Pantoprazole Sodium 40 mg DR Tablet (test) dosed in first period followed by Protonix® 40 mg DR Tablet (reference) dosed in second period
- Protonix® (Reference) First: Protonix 40 mg DR Tablet (reference) dosed in first period followed by Pantoprazole Sodium 40 mg DR Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Pantoprazole (Test) First | Protonix® (Reference) First
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0
Period: Washout: 5 Days
Arm/Group | Pantoprazole (Test) First | Protonix® (Reference) First
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Pantoprazole (Test) First | Protonix® (Reference) First
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pantoprazole (Test) First | Protonix® (Reference) First | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 31 | 36 | 67
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 41 | 42 | 83
  Black | 5 | 5 | 10
  American Indian | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Hispanic | 2 | 1 | 3
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration - Pantoprazole in Plasma
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 16 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Pantoprazole: Pantoprazole Sodium 40 mg DR Tablet (test) dosed in either period
- Protonix®: Protonix 40 mg DR Tablet (reference) dosed in either period
Arm/Group | Pantoprazole | Protonix®
Number analyzed (Participants) | 100 | 100
ng/mL | 2494.120 (965.022) | 2747.380 (879.942)
Statistical Analysis 1: Comparison: Pantoprazole vs Protonix®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 88.8, 90% CI [82.7 to 95.4] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 16 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis. Not all subjects data could be used to estimate AUC0-inf.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Pantoprazole | Protonix®
Number analyzed (Participants) | 96 | 99
ng*h/mL | 6280.022 (6311.033) | 6332.279 (5923.458)
Statistical Analysis 1: Comparison: Pantoprazole vs Protonix®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 97.3, 90% CI [93.4 to 101] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 16 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Pantoprazole | Protonix®
Number analyzed (Participants) | 100 | 100
ng*h/mL | 5822.470 (4825.928) | 6016.176 (4502.333)
Statistical Analysis 1: Comparison: Pantoprazole vs Protonix®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 95.6, 90% CI [91.6 to 99.8] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.